CLINICAL TRIAL: NCT02011022
Title: Pharmacokinetic Analysis of High Dose Methotrexate in Pediatric Acute Lymphoblastic Leukemia: Significant Impact Factors and Establishment of a Clinically Relevant Model
Brief Title: Pharmacokinetic Analysis of High Dose Methotrexate in Pediatric Lymphoblastic Malignancies
Acronym: HDMTX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Weiqun Xu, Doctor, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: chzj-HDMTX-20131205
Record Dates: First submitted 2013-12-05; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Methotrexate Adverse Reaction
Keywords: Methotrexate,; Pharmacokinetic; Acute lymphoblastic leukemia; Model
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3g group (Experimental): The dose of MTX is 3 g/m2
  Interventions: Drug: 3g MTX
- 5g group (Experimental): The dose of MTX is 5g/m2
  Interventions: Drug: 5g MTX

INTERVENTIONS:
Drug: 3g MTX — The group of patients which are treated with 3g/m2 MTX, low risk ALL or NHL
  Arms: 3g group
Drug: 5g MTX — The group of patients which are treated with 5g/m2 MTX, they are high or middle risk ALL patients
  Arms: 5g group

SUMMARY:
* The pharmacokinetics of MTX were assessed with regards to the relevance of several different patient specific factors in 291 pediatric patients, who were administered with high dose of MTX. Population pharmacokinetics of MTX analysis was performed by using nonlinear mixed effects modeling.

DETAILED DESCRIPTION:
* Methotrexate (MTX) is one of the critical components for treating all forms of acute lymphoblastic leukemia (ALL), which is the most common pediatric cancer. Unfortunately, high dose MTX has several undesirable side effects and MTX toxicity vastly differs from patient to patient.
* The pharmacokinetics of MTX were assessed with regards to the relevance of several different patient specific factors in 291 pediatric patients, who were administered with high dose of MTX. Population pharmacokinetics of MTX analysis was performed by using nonlinear mixed effects modeling.
* The final model was validated using nonparametric bootstrap analysis. Body surface area (BSA), pre-hydration, baseline serum creatinine and 24 h creatinine clearance rate were statistically significant covariates for distributional volume (V) and renal clearance (CL). Herein, is the first report of analysis of the importance of a series of patient factors on pharmacokinetics of MTX by one-compartment model. Using these data, we have established an efficient population pharmacokinetic model for MTX, which can be used to predict safe clinical application of MTX especially in children with ALL.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia and non-hodgkin's lymphoma younger than 18 years old

Exclusion Criteria:

* Non lymphoblastic malignancies or older than 18 years

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 291 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
elimination delay | 3 days
  The serum MTX is higher than 1umol/L in 48 hours or 0.1umol/L in 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Weiqun Xu, Principal Investigator — The Children's Hospital of Zhejiang University School of Medicine
Locations (1):
- The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Yanagimachi M, Goto H, Kaneko T, Naruto T, Sasaki K, Takeuchi M, Tanoshima R, Kato H, Yokosuka T, Kajiwara R, Fujii H, Tanaka F, Goto S, Takahashi H, Mori M, Kai S, Yokota S. Influence of pre-hydration and pharmacogenetics on plasma methotrexate concentration and renal dysfunction following high-dose methotrexate therapy. Int J Hematol. 2013 Dec;98(6):702-7. doi: 10.1007/s12185-013-1464-z. Epub 2013 Nov 16. PMID 24241962
- See also: Another related article — http://www.ncbi.nlm.nih.gov/pubmed/24158402